CLINICAL TRIAL: NCT03323164
Title: Changes in Peripapillary Blood Flow After Use of Anti-glaucoma Medications: A Prospective, Quantitative OCT Angiography Study
Brief Title: Peripapillary Blood Flow After Use of Anti-glaucoma Medications: An OCT Angiography Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Optovue (Industry)
Responsible Party: Principal Investigator, Daniel Lee, MD, Principal Investigator, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17-636E
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Glaucoma; Drugs; Normal Tension Glaucoma; Primary Open-angle Glaucoma
MeSH Terms: conditions — Glaucoma; Low Tension Glaucoma; Glaucoma, Open-Angle | interventions — Timolol; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Timolol (Active Comparator): Timolol maleate 0.5% ophthalmic solution Instillation of one drop in each eye, once.
  Interventions: Drug: Timolol Maleate
- Brimonidine (Active Comparator): Brimonidine tartrate 0.2% Instillation of one drop in each eye, once.
  Interventions: Drug: Brimonidine Tartrate

INTERVENTIONS:
Drug: Timolol Maleate — Instillation of one drop in each eye, one-time. Obtaining of OCT angiography scans after 2 hours of instillation.
  Other Names: Timolol
  Arms: Timolol
Drug: Brimonidine Tartrate — Instillation of one drop in each eye, one-time. Obtaining of OCT angiography scans after 2 hours of instillation.
  Other Names: Brimonidine
  Arms: Brimonidine

SUMMARY:
This study evaluates the possible acute changes in peripapillary blood flow after instillation of antiglaucoma medications in patients with primary open angle glaucoma (POAG), normal tension glaucoma (NTG), or ocular hypertension (OHTN) using Optical Coherence Tomography (OCT) angiography.

DETAILED DESCRIPTION:
Reduction of intraocular pressure (IOP) with topical antihypertensive medications is the mainstay of initial treatment in patients with OHTN, POAG, and NTG. Many patients, however, continue to experience disease progression despite IOP reduction. Alternative mechanisms of neurodegeneration, including vascular dysregulation and structural susceptibility of the lamina cribrosa, have been proposed as important mechanisms in progression, particularly in cases of NTG.

Prior studies have also found decreased calculated mean ocular perfusion with the use of timolol compared to other antiglaucoma medications in patients with normal tension glaucoma. Visual field deterioration has also been shown to be associated with systemic nocturnal arterial hypotension in patients with NTG, POAG, and after anterior ischemic optic neuropathy. The use of ophthalmic topical beta-blockers has been shown to lower nocturnal diastolic blood pressure and heart rate. Thus, topical beta blockers are often avoided in the treatment of NTG due to the potential risk of reduced optic nerve head perfusion

Studies evaluating optic nerve head (ONH) perfusion are limited. Earlier studies evaluated indirect measurements, such as calculated mean ocular perfusion pressure or systemic hypotension, as indications of optic nerve hypoperfusion. Direct measurements of ocular perfusion have been attempted using retrobulbar color Doppler imaging, which demonstrated decreased short posterior ciliary artery flow velocity in patients with glaucomatous visual field progression. This technique, however, has yielded inconsistent results in other studies, and is only capable of detecting gross changes to ocular blood flow.

Optical Coherence Tomography Angiography (OCTA) is a novel technique first introduced in 2014 using a custom swept-source OCT system.No studies currently exist to evaluate the effects of antiglaucoma medications on peripapillary blood flow using OCTA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ocular hypertension, primary open angle glaucoma, or normal tension glaucoma in the study eye(s)
* Age 18-90
* Best corrected visual acuity of 20/60 or better

Exclusion Criteria:

* Current use of either brimonidine or timolol
* Other disease, ophthalmic or systemic, that is likely to significantly affect the OCT test in the study eye(s) including:

  * More than moderate grade cataract that significantly reducing OCTA scan signal level
  * Macular degeneration other than mild drusen or pigmentary changes
  * Diabetic retinopathy other than mild background non proliferative retinopathy
  * Prior or current macular edema
  * Prior laser treatment to the retina
  * Prior retinal detachment
  * Prior central serous retinopathy
  * Prior retinal vein or artery occlusion
  * Prior inflammatory retinopathy or choroidopathy
  * Keratoconus or other corneal ectasia
  * Corneal scarring in central 4 mm
  * Prior penetrating keratoplasty
  * Ischemic optic neuropathy
  * Dementia beyond early/mild memory loss
  * History of cerebrovascular accident
  * History of severe carotid stenosis
  * History of previous ocular surgery other than non-complicated cataract extraction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lee, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Glaucoma Research Center - Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Timolol: Timolol maleate 0.5% ophthalmic solution Instillation of one drop in each eye, once.
  Timolol Maleate: Instillation of one drop in each eye, one-time. Obtaining optical coherence tomography (OCT) angiography scans after 2 hours of instillation.
- Brimonidine: Brimonidine tartrate 0.2% Instillation of one drop in each eye, once.
  Brimonidine Tartrate: Instillation of one drop in each eye, one-time. Obtaining optical coherence tomography (OCT) angiography scans after 2 hours of instillation.
Period: Overall Study
Arm/Group | Timolol | Brimonidine
Started | 18 | 17
Completed | 16 | 15
Not Completed | 2 | 2
Not completed — Poor quality imaging/scans | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Timolol | Brimonidine | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 13 | 29
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 13 | 8 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31
Glaucoma type [Count of Participants; unit: Participants] — Patients diagnosed with primary open angle glaucoma (POAG), normal tension glaucoma (NTG) or ocular hypertension (OHTN), with a best corrected visual acuity of at least 20/60 were invited to participate.
  Participants | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Changes in Vessel Density in Treatment Groups Assessed by OCT Angiography
Description: Percent change in peripapillary vessel density detected by OCT (optical coherence tomography) Angiography using spectrum amplitude decorrelation angiography (SSADA) algorithm with the use of topical brimonidine or timolol eye drops to lower eye pressure.
Time Frame: 5.5 hours (3 separate 30 minute OCT Angiography scans with 2 hour post-intervention in between each scan)
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Brimonidine Group: POAG (primary open angle glaucoma), NTG (normal tension glaucoma) and OHTN (ocular hypertension) had OCTA (optical coherence tomography angiography) after receiving Brimonidine eye drops to lower eye pressure before .
- Timolol Group: POAG (primary open angle glaucoma), NTG (normal tension glaucoma) and OHTN (ocular hypertension) had OCTA (optical coherence tomography angiography) after receiving Timolol eye drops to lower eye pressure before .
Arm/Group | Brimonidine Group | Timolol Group
Number analyzed (Participants) | 15 | 16
percent change
  Overall group | -0.51 (6.10) | 2.59 (6.47)
  POAG | -0.96 (8.069) | 0.96 (6.71)
  NTG | -0.04 (6.67) | 4.12 (8.11)
  OHTN | -0.58 (4.48) | 2.37 (4.77)

2. Primary Outcome: Changes in Flow Index in Treatment Groups Assessed by OCT Angiography
Description: Percent change in peripapillary Flow Index detected by OCT (optical coherence tomography) Angiography using spectrum amplitude decorrelation angiography (SSADA) algorithm with the use of topical brimonidine or timolol eye drops to lower eye pressure.
Time Frame: 5.5 hours (3 separate 30 minute OCT Angiography scans with 2 hour post-intervention in between each scan)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Brimonidine Group | Timolol Group
Number analyzed (Participants) | 15 | 16
percent change
  Overall group | -5.23 (10.77) | 0.33 (5.11)
  POAG | -12.55 (12.01) | 0.69 (7.64)
  NTG | -4.87 (6.35) | 2.76 (2.55)
  OHTN | 1.71 (9.68) | -2.92 (3.05)

3. Primary Outcome: Comparison of Percent Changes in Peripapillary Vessel Density in Treatment Groups Assessed by OCT Angiography
Description: Comparison of the percent change in peripapillary vessel density detected by OCT (optical coherence tomography) Angiography using spectrum amplitude decorrelation angiography (SSADA) algorithm before and after the use of topical brimonidine or timolol eye drops to lower eye pressure. The Control groups represent the percent changes in vessel density after using artificial tears. The medicine groups (Brimonidine/Timolol) represents the percent changes in vessel density after using topical brimonidine or timolol drops to lower eye pressure.
Time Frame: 5.5 hours (3 separate 30 minute OCT Angiography scans with 2 hour post-intervention in between each scan)
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Control B: POAG (primary open angle glaucoma), NTG (normal tension glaucoma) and OHTN (ocular hypertension) had OCTA (optical coherence tomography angiography) before receiving Brimonidine eye drops to lower eye pressure before .
- Brimonidine: POAG (primary open angle glaucoma), NTG (normal tension glaucoma) and OHTN (ocular hypertension) had OCTA (optical coherence tomography angiography) after receiving Brimonidine eye drops to lower eye pressure before .
- Control T: POAG (primary open angle glaucoma), NTG (normal tension glaucoma) and OHTN (ocular hypertension) had OCTA (optical coherence tomography angiography) before receiving Timolol eye drops to lower eye pressure before .
- Timolol: POAG (primary open angle glaucoma), NTG (normal tension glaucoma) and OHTN (ocular hypertension) had OCTA (optical coherence tomography angiography) after receiving Timolol eye drops to lower eye pressure before .
Arm/Group | Control B | Brimonidine | Control T | Timolol
Number analyzed (Participants) | 15 | 15 | 16 | 16
percent change
  Overall group | 1.70 (6.68) | -0.51 (6.10) | -2.05 (3.90) | 2.59 (6.47)
  POAG | 2.89 (10.73) | -1.62 (9.15) | -2.8 (4.64) | 0.96 (6.71)
  NTG | 2.02 (5.59) | -0.04 (6.67) | -3.42 (4.01) | 4.12 (8.11)
  OHTN | 0.44 (4.89) | -0.58 (4.48) | 0.34 (2.21) | 2.37 (4.77)

4. Primary Outcome: Comparison of Percent Changes in Peripapillary Flow Index in Treatment Groups Assessed by OCT Angiography
Description: Comparison of the percent change in peripapillary flow index detected by OCT (optical coherence tomography) Angiography using spectrum amplitude decorrelation angiography (SSADA) algorithm before and after the use of topical brimonidine or timolol eye drops to lower eye pressure. The Control groups represent the percent changes in flow index after using artificial tears. The medicine groups (Brimonidine/Timolol) represents the percent changes in flow index after using topical brimonidine or timolol drops to lower eye pressure.
Time Frame: 5.5 hours (3 separate 30 minute OCT Angiography scans with 2 hour post-intervention in between each scan)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Control B | Brimonidine | Control T | Timolol
Number analyzed (Participants) | 15 | 15 | 16 | 16
percent change
  Overall group | 2.35 (11.66) | -5.23 (10.77) | 1.61 (11.10) | 0.33 (5.11)
  POAG | 12.81 (15.26) | -14.91 (12.45) | -3.65 (5.33) | 0.69 (7.64)
  NTG | 0.22 (1.95) | -4.87 (6.35) | 7.57 (16.31) | 2.76 (2.55)
  OHTN | -3.89 (9.97) | 1.71 (9.68) | -0.26 (2.95) | -2.92 (3.05)

5. Primary Outcome: Comparison of Percent Changes in Optic Nerve Head Vessel Density in Treatment Groups Assessed by OCT Angiography
Description: Comparison of the percent change in optic nerve head vessel density detected by OCT (optical coherence tomography) Angiography using spectrum amplitude decorrelation angiography (SSADA) algorithm before and after the use of topical brimonidine or timolol eye drops to lower eye pressure. The Control groups represent the percent changes in vessel density after using artificial tears. The medicine groups (Brimonidine/Timolol) represents the percent changes in vessel density after using topical brimonidine or timolol drops to lower eye pressure.
Time Frame: 5.5 hours (3 separate 30 minute OCT Angiography scans with 2 hour post-intervention in between each scan)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Control B | Brimonidine | Control T | Timolol
Number analyzed (Participants) | 15 | 15 | 16 | 16
Percent change
  Overall | 1.27 (6.95) | 1.08 (6.67) | 0.32 (4.96) | 0.91 (5.45)
  POAG | 2.22 (7.87) | -1.00 (6.02) | -2.68 (4.37) | 2.65 (4.89)
  NTG | 2.13 (7.03) | 2.44 (8.21) | 1.70 (6.30) | 0.16 (7.40)
  OHTN | -0.34 (7.50) | 1.65 (7.31) | 1.67 (2.66) | 0.08 (3.66)

6. Primary Outcome: Comparison of Percent Changes in Optic Nerve Head Flow Index in Treatment Groups Assessed by OCT Angiography
Description: Comparison of the percent change in Optic Nerve Head Flow Index detected by OCT (optical coherence tomography) Angiography using spectrum amplitude decorrelation angiography (SSADA) algorithm before and after the use of topical brimonidine or timolol eye drops to lower eye pressure. The Control groups represent the percent changes in flow index after using artificial tears. The medicine groups (Brimonidine/Timolol) represents the percent changes in flow index after using topical brimonidine or timolol drops to lower eye pressure.
Time Frame: 5.5 hours (3 separate 30 minute OCT Angiography scans with 2 hour post-intervention in between each scan)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Control B | Brimonidine | Control T | Timolol
Number analyzed (Participants) | 15 | 15 | 16 | 16
percent change
  Overall | 2.69 (12.08) | -5.24 (10.05) | 1.96 (9.08) | -0.69 (5.37)
  POAG | 12.40 (14.22) | -13.73 (11.02) | -2.38 (3.64) | -1.65 (7.54)
  NTG | 0.32 (3.42) | -4.17 (5.77) | 6.21 (13.79) | 2.47 (2.65)
  OHTN | -2.68 (13.18) | 0.55 (10.65) | 1.21 (2.61) | -3.52 (4.04)

ADVERSE EVENTS:
Time Frame: 4 hours
Arm/Group | Timolol | Brimonidine
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

LIMITATIONS AND CAVEATS:
Limited sample size in this pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT03323164/Prot_SAP_000.pdf